CLINICAL TRIAL: NCT00537589
Title: Randomized Control Trial of Ultrasound-Guided Peripheral Arthrocentesis
Brief Title: Ultrasound Guided Arthrocentesis
Acronym: UGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-04-06A
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2007-09

CONDITIONS: Arthritis; Joint Pain
Keywords: arthrocentesis; ultrasound; emergency
MeSH Terms: conditions — Arthritis; Arthralgia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ultrasound guided arthrocentesis — Guidance of joint aspiration by ultrasound guidance

SUMMARY:
Does ultrasound guidance improve success rate and decrease aspiration attempts for peripheral arthrocentesis?

ELIGIBILITY:
Inclusion Criteria:

* Age at or over 18
* Indication for peripheral arthrocentesis

Exclusion Criteria:

* Hemodynamic instability
* Previous arthroplasty of the joint
* Known intraarticular fracture
* Hip arthrocentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2004-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Success rate for arthrocentesis | within ED visit

SECONDARY OUTCOMES:
Reduction in aspiration attempts | within ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Vivek S Tayal, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States